CLINICAL TRIAL: NCT03320317
Title: BIC4CRC: Breakthrough Improvement Collaborative for ColoRectal Cancer
Brief Title: Breakthrough Improvement Collaborative for ColoRectal Cancer (BIC4CRC)
Acronym: BIC4CRC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Principal Investigator, Kris Vanhaecht, Professor, KU Leuven
Other Study IDs: BIC4CRC/2017/1
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal cancer
  Interventions: Other: Learning session 1; Other: Learning session 2; Other: Learning session 3; Other: Learning session 4

INTERVENTIONS:
Other: Learning session 1 — Learn form international report, Explain key interventions, Explain BIC methodology, Retrospective patient record analysis, Team measures
Other: Learning session 2 — Feedback report, Share (inter)national best practices, Discussion, set priorities, teaching and improvement, Retrospective patient record analysis
Other: Learning session 3 — Feedback report, Share best practices, Discussion, set priorities, teaching and improvement, Retrospective patient record analysis, Team measures
Other: Learning session 4 — Feedback report, Best practice symposium

SUMMARY:
Colorectal cancer is the most common cancer in Europe and the third worldwide. Approximately 1 in 20 men and 1 in 35 women will develop colorectal cancer at some moment in their life. In Flanders, in 2014, there was an increase in the detection of colorectal cancer with 21% compared to 2013. Early detection improves the prognosis for the patient. In this early stage, colorectal surgery is one of the most important treatments, but it is also complex and has a high complication rate. However, over the last decade, surgical care for patients with colorectal cancer has become more standardized. The use of structured care methods, such as care pathways and protocols, has helped in standardizing care processes. Specifically for patients with colorectal cancer, perioperative care has shifted with the implementation of Enhanced Recovery After Surgery (ERAS) programs. The goal of ERAS- protocols is to optimize the interventions during the perioperative hospitalization period and reduce postoperative complications. Despite the increasing evidence in favor of the use of these standardized protocols, adherence and implementation in daily practice remains challenging.

The primary goal of this quality improvement project is to enhance the standardization of key interventions in the ERAS care process for patients undergoing colorectal surgery.

Therefore, adherence to the ERAS-guidelines will be investigated and hospitals will receive feedback to set up improvement initiatives. Moreover, interactive group sessions and on-site training activities will stimulate knowledge sharing and define best practices.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Elective admission for colorectal cancer surgery

Exclusion Criteria:

* Emergency (not planned) admission for colorectal cancer surgery
* Patients diagnosed with severe dementia or severe concomitant disease that may affect very short term outcome and hence influence deviations from standard acute care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with colorectal cancer admitted for planned surgery
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of stay | through study completion, an average of 4 months
  Number of days in the hospital

SECONDARY OUTCOMES:
30-days readmission rate | through study completion, an average of 4 months
  Readmission rate
Mortality rate | through study completion, an average of 4 months
  Mortality rate
Complication rate | through study completion, an average of 4 months
  Re-intervention, wound complications, surgical site infection, anastomotic leak or stoma related complications

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-brabant, Belgium

REFERENCES:
- [Background] van Zelm R, Janssen I, Vanhaecht K, de Buck van Overstraeten A, Panella M, Sermeus W, Coeckelberghs E. Development of a model care pathway for adults undergoing colorectal cancer surgery: Evidence-based key interventions and indicators. J Eval Clin Pract. 2018 Feb;24(1):232-239. doi: 10.1111/jep.12700. Epub 2017 Feb 1. PMID 28145019
- [Background] van Zelm R, Coeckelberghs E, Sermeus W, De Buck van Overstraeten A, Weimann A, Seys D, Panella M, Vanhaecht K. Variation in care for surgical patients with colorectal cancer: protocol adherence in 12 European hospitals. Int J Colorectal Dis. 2017 Oct;32(10):1471-1478. doi: 10.1007/s00384-017-2863-z. Epub 2017 Jul 17. PMID 28717841